CLINICAL TRIAL: NCT03442712
Title: Feasibility of Self-administered Auricular Acupressure Integrated With Mobile Device Reminders for Weight Reduction.
Brief Title: Auricular Acupressure Integrated With Mobile Device for Weight Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Lorna Suen, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UADZ
Record Dates: First submitted 2018-02-12; First posted 2018-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Weight Loss; Mobile Application; Ear Acupressure
Keywords: obesity; weight loss; ear acupressure; smartphone application
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Intervention Model Description: This study is a three-arm randomised waitlist-controlled feasibility trial.
Who Masked: Outcomes Assessor
Masking Description: The effects of the treatment will be evaluated by another researcher (second RA) who is blinded to the type of treatment modality received by the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment arm 1 (Active Comparator): Auricular acupressure (AA) plus smartphone App:
  Semen Vaccaria laccaria will be applied on one ear only, and seed plasters will be changed every 3 days to 4 days to the opposite ear. Subjects will be requested to apply pressure on the acupoints thrice per day. The subjects will install the smartphone App specifically designed for this study. The App will send out regular AA reminders to the subjects. The total treatment period will be 8 weeks.
  Interventions: Other: Auricular acupressure plus smartphone App
- Treatment arm 2 (Active Comparator): The participants will only receive AA treatment and are required to perform daily self-administered seeds pressing.
  Interventions: Other: Auricular acupressure
- Treatment arm 3 (No Intervention): The participants in the waitlist control group will maintain their usual dietary and exercising patterns.

INTERVENTIONS:
Other: Auricular acupressure plus smartphone App — Semen Vaccaria laccaria will be kept in place by a piece of adhesive patch. Seeds will be applied on one ear only, and seed plasters will be changed every 3 days to 4 days to the opposite ear, that is, we will meet the subjects twice per week. Subjects will be requested to apply pressure on the acupoints thrice per day, preferably within 30 min before eating, pressing for 20 times using a constant rhythm to each point. Coaching on how to self-administer AA on the acupoints will be given to the subjects, and a return demonstration from the subjects will be required to ensure the skills are performed properly. The subjects will install the smartphone App specifically designed for this study. The App will send out regular AA reminders to the subjects. In addition, the subjects will be asked to input the number of bowel open and compliance with AA performance per day into the App. The total treatment period will be 8 weeks.
  Arms: Treatment arm 1
Other: Auricular acupressure — The participants will receive AA treatment and are required to perform daily self-administered seeds pressing, but no smartphone App will be provided, but a booklet containing relevant information will be provided to the subjects.
  Arms: Treatment arm 2

SUMMARY:
Obesity is a common global health problem. A three-arm randomised waitlist-controlled feasibility trial is proposed. A total of 59 subjects (19-21 subjects per arm) will be recruited. The three groups are AA plus smartphone application (experimental group); AA only (comparison group); and Waitlist control group. In the experimental group, seeds will be applied on six specific ear acupoints of the subjects by the researcher. Subjects will be requested to apply pressure on the acupoints thrice per day. They will install a smartphone App which will send out regular reminders for pressing, allow the subjects to input the number of bowel open, compliance rate, and difficulties entered during the process for timely advice. The total treatment period will be 8 weeks. Outcome measures will be conducted at baseline and postintervention at 8 weeks, including obesity and anthropometric index, leptin concentration and adiponectin level. Patient satisfaction towards the therapy, the use of the smartphone application and the implementation of the treatment protocol will be determined.

DETAILED DESCRIPTION:
Obesity is a common global health problem. It increases the risk of many chronic illnesses, such as hypertension, type 2 diabetes mellitus and cardiovascular diseases. Conventional approaches to alleviate obesity are medications, exercise, dietary control, behaviour modification therapy or bariatric surgeries. However, the safety of anti-obesity agents is a concern, and gastric bypass surgery and other bariatric surgeries also pose potential risks after operation. Auricular acupuncture therapy is frequently used to treat obesity. However, the use of needles for auricular acupuncture may be unacceptable to people. Some researchers attempted to adopt a combined approach by integrating auriculotherapy with diet restriction, and the effect solely attributed to auriculotherapy cannot be determined. On the other hand, auricular acupressure (AA) is a safe, noninvasive, inexpensive and easily self-administered approach that causes very few adverse effects. Previous evidence has demonstrated that AA is an effective intervention to reduce body weight, increase satiety and self-efficacy on weight control through the self-administration of seeds pressing several times per day, after the seeds are applied by the researchers on the ear acupoints. It is associated with the decreased leptin levels and an increase of adiponectin level in which these hormones are associated with weight loss. However, therapists may have difficulties to monitor the compliance of subjects to perform seed pressing which in turn affecting the intervention dosages. This study aims to evaluate the feasibility of self-administered AA integrated with mobile device reminders for weight reduction in individuals with overweightness or obesity. A three-arm randomised waitlist-controlled feasibility trial is proposed. A total of 59 subjects (19-21 subjects per arm) will be recruited. The three groups are AA plus smartphone application (experimental group); AA only (comparison group); and Waitlist control group. In the experimental group, seeds will be applied on six specific ear acupoints of the subjects by the researcher. Subjects will be requested to apply pressure on the acupoints thrice per day. They will install a smartphone App which will send out regular reminders for pressing, allow the subjects to input the number of bowel open, compliance rate, and difficulties entered during the process for timely advice. The total treatment period will be 8 weeks. Outcome measures will be conducted at baseline and postintervention at 8 weeks, including obesity and anthropometric index, leptin concentration and adiponectin level. Patient satisfaction towards the therapy, the use of the smartphone application and the implementation of the treatment protocol will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Overweightness, with body mass index (BMI) ≥ 25.0 kg/m2 in accordance with the BMI classification of the World Health Organization (WHO)
* Subjects that have neither received other weight control measures (manoeuvres) nor experienced medical and/or drug history within the last 3 months
* No ear injury, such as inflammation or lesions, and no medical history of ear surgery within the last 6 months
* Smartphone user (IOS and android)

Exclusion criteria:

(1) diabetes, severe hypertension, heart disease or endocrine abnormalities,; (2) pregnancy; (3) eating disorders screened with a 5-item SCOFF questionnaire (Bradford et al. 2010); (4) psychiatric and mental disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
body mass index | up to 8 weeks
  body mass index is defined as the body mass divided by the square of the body height, i.e. kg/meter square

SECONDARY OUTCOMES:
Appetite parameters which include hunger, fullness and satiety level | up to 8 weeks
  Participants will be asked to compete the Visual Analogue Scale (VAS) before lunch and dinner meals taking an average for three consecutive days at each timepoints (baseline, and post-intervention at 8 weeks), using VAS scale to measure the appetite in terms of hunger, fullness and satiety level.
Leptin concentration | up to 8 weeks
  leptin concentration will be measured in duplicate by using a commercial sandwich ELISA kit comprising ready-to-use components, which are either concentrated or lyophilised.
Adiponectin level | up to 8 weeks
  Adiponectin level will be measured with a commercially available sandwich ELISA kit
Participants' expectation | baseline
  A 5-item participants' expectation questionnaire will be collected from the participants.
Patient satisfaction | up to 8 weeks
  Patient satisfaction towards the therapy, the use of the smartphone app and the implementation of the treatment protocol will be determined.
Bowel open | up to 8 weeks
  bowel open per day
Fat percentage | up to 8 weeks
  this include body fat percentage, visceral fat level, and segmental subcutaneous fat percentage
waist hip ratio | up to 8 weeks
  It is the dimensionless ratio of the circumference of the waist to that of the hips, calculated as waist measurement divided by hip measurement

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Suen, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Suen L, Wang W, Cheng KKY, Chua MCH, Yeung JWF, Koh WK, Yeung SKW, Ho JYS. Self-Administered Auricular Acupressure Integrated With a Smartphone App for Weight Reduction: Randomized Feasibility Trial. JMIR Mhealth Uhealth. 2019 May 29;7(5):e14386. doi: 10.2196/14386. PMID 31144666